CLINICAL TRIAL: NCT01529606
Title: Development of a Miniature Plasma Brush for Dental Clinical Applications
Brief Title: Cold Plasma for Dental Restoration and Caries Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanova, Inc (Industry)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Liang Hong, Associate Professor and Director, University of Tennessee
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R44DE019041 (NIH); 5R44DE019041 (NIH)
Record Dates: First submitted 2012-02-03; First posted 2012-02-09 (Estimated); Results first posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Dental Restoration; Caries
Keywords: dental restoration; dental caries; tooth cavity
MeSH Terms: conditions — Dental Caries | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care (Active Comparator): Fifty patients will be recruited into standard treatment group and they will receive composite resin restoration for all decayed teeth and standard preventive treatment (cleaning and fluoride varnish application) at baseline.
  Interventions: Other: Composite restoration and tooth cleaning
- Plasma treatment (Experimental): Fifty patients will be recruited into plasma treatment group and they will receive plasma treatment after cavity preparation, composite resin restoration, standard preventive treatment followed by plasma treatment for non-carious teeth.
  Interventions: Procedure: Plasma treatment

INTERVENTIONS:
Other: Composite restoration and tooth cleaning — Standard preventive treatment will be repeated on semi-annual (6-month) recall visits. All composite restorations will be placed according to the manufacturer's instruction.
  Other Names: Standard composite filling and preventive treatment
  Arms: Standard care
Procedure: Plasma treatment — plasma treatment after preparation and for caries prevention
  Other Names: Plasma treatment and standard preventive treatment
  Arms: Plasma treatment

SUMMARY:
The main objective of this entire research project is to develop a miniature atmospheric cold plasma brush (m-ACPB) for dental clinical applications. The objective of the clinical trial portion of the study is to compare the longevity and durability of dental composite restorations created using the plasma brush, to that of the standard care in dentistry for treating dental cavities, and effects on caries prevention.

DETAILED DESCRIPTION:
The study will be a randomized controlled trial (RCT) and be approved by the institute review board of the University of Tennessee Health Science Center. The study subjects will be composed of young adults 18-35 years old in order to control effects of age on caries. Also the subjects must be Caucasian or Africa American. Young adult patients will be recruited from the UTHSC dental clinics.The baseline visit include a dental exam by one of the investigators, standard preventive dental care (e.g cleaning, application of fluoride varnish), anthropometric measurements, oral health interview survey. 100 patients who meet all inclusion and exclusion criteria will be recruited after they sign an informed consent form. These patients will be randomly assigned to 1 of 2 study groups. Randomization assignment will be stratified by age and number of teeth with caries. Two study groups will be: 1.) plasma treatment group and 2) standard treatment group. For patients in standard treatment group, they will receive composite resin restoration for all decayed teeth and standard preventive treatment (cleaning and fluoride varnish application) at baseline. For patients in plasma treatment group, they will receive plasma treatment after cavity preparation, composite resin restoration, standard preventive treatment followed by plasma treatment for non-carious teeth. Standard preventive treatment and plasma treatment will be repeated on semi-annual (6-month) recall visits. All composite restorations will be placed according to the manufacturer's instruction. Only one composite commercially available will be used during the study.

ELIGIBILITY:
Inclusion Criteria:

* subject must be Caucasian or Africa American, 18-35 years old, have written, completed, informed consent forms;
* be generally healthy;
* be able to participate in the study;
* have no diagnosed periodontitis and pericoronitis;
* have no active mucosal diseases such as aphthous ulcers and herpetic stomatitis.

They must also agree to follow study instructions.

The patients must meet the following specific entry criteria:

* 1-5 untreated caries and at least one class II caries.

Exclusion Criteria:

* each subject must have no diagnosed diabetes mellitus or any other endocrine diseases;
* no diagnosed cardiovascular diseases;
* no diagnosed immune-compromised diseases, such as HIV and AIDS;
* no other serious systemic diseases, such as cancer;
* no antibiotic therapy in the past 6 months;
* no use of non-steroidal anti-inflammatory drugs (NSAIDS) in the past 3 months; and
* no reported use of illicit drugs.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2012-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liang Hong, DDS, Ph.D, Principal Investigator — The University of Tennessee Health Science Center
Locations (1):
- University of Tennessee Health Science, Memphis, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two more patients were recruited because patients received recruitment information and requested participation in the study.
Period: Overall Study
Arm/Group | Standard Care | Plasma Treatment
Started | 55 | 47
Completed | 34 | 29
Not Completed | 21 | 18
Not completed — Lost to Follow-up | 21 | 18

BASELINE CHARACTERISTICS:
Groups:
- Standard Care: Fifty five patients were recruited into standard treatment group and they will receive composite resin restoration for all decayed teeth and standard preventive treatment (cleaning and fluoride varnish application) at baseline.
  Composite restoration and tooth cleaning: Standard preventive treatment will be repeated on semi-annual (6-month) recall visits. All composite restorations will be placed according to the manufacturer's instruction.
- Plasma Treatment: Forty seven patients were recruited into plasma treatment group and they will receive plasma treatment after cavity preparation, composite resin restoration, standard preventive treatment followed by plasma treatment for non-carious teeth.
  Plasma treatment: plasma treatment after preparation and for caries prevention
- Total: Total of all reporting groups
Arm/Group | Standard Care | Plasma Treatment | Total
Number analyzed (Participants) | 55 | 47 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 47 | 102
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.9 (4.4) | 27.7 (4.6) | 27.8 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 32 | 67
  Male | 20 | 15 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 39 | 27 | 66
  White | 16 | 20 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 55 | 47 | 102
Education level [Count of Participants; unit: Participants]
  High school or below | 10 | 8 | 18
  Some college | 18 | 11 | 29
  4 year college | 8 | 12 | 20
  Graduate or professional school | 19 | 16 | 35
Income level [Count of Participants; unit: Participants]
  <$20,000 | 23 | 22 | 45
  $20,000-$39,999 | 21 | 19 | 40
  $40,000-$59,999 | 2 | 5 | 7
  $60,000 or more | 9 | 1 | 10
Health Insurance [Count of Participants; unit: Participants]
  Yes | 42 | 30 | 72
  No | 13 | 17 | 30
Tooth brushing [Count of Participants; unit: Participants]
  >=3 times per day | 8 | 5 | 13
  Twice per day | 31 | 32 | 63
  Once per day | 13 | 10 | 23
  <one time per day | 3 | 0 | 3
Number of decayed, missing and filling teeth [Mean (Standard Deviation); unit: tooth] | 6.09 (4.22) | 5.00 (4.55) | 5.54 (4.38)
Number of decayed and filling surfaces (DMFS) [Mean (Standard Deviation); unit: tooth surface] | 8.27 (8.28) | 6.89 (7.50) | 7.58 (7.76)
Number of decayed surfaces (DS) [Mean (Standard Deviation); unit: tooth surface] | 2.06 (6.57) | 0.66 (1.73) | 1.57 (3.48)

OUTCOME MEASURES:

1. Primary Outcome: Number of Decayed, Missing and Filling Teeth (DMFT)
Description: Number of decayed, missing and filling teeth (DMFT) during 12 months
Time Frame: 12 months
Population: 34 participants in standard care group and 29 in plasma group
Measure: Mean (Standard Deviation); unit: teeth
Arm/Group | Standard Care | Plasma Treatment
Number analyzed (Participants) | 34 | 29
teeth | 6.29 (4.07) | 5.14 (4.70)

2. Primary Outcome: Decayed and Filling Surfaces
Description: Number of decayed and filling surfaces
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: tooth surface
Arm/Group | Standard Care | Plasma Treatment
Number analyzed (Participants) | 34 | 29
tooth surface | 9.03 (8.14) | 7.72 (8.16)

3. Primary Outcome: Restoration Failure Rate
Description: Composite restoration evaluation for fracture or loss of filling partially or completely, with or without recurrent caries.
Time Frame: 12 months
Population: After 12 months, in standard care group, we had 27 participants remaining and lost 28 participants; in plasma treatment group, we had 21 participants remaining and lost 26 participants. Units of analysis for composite restoration failure is number of composite restorations in each group. A participant may have more than one composite restoration.
Measure: Number; unit: composite fillings
Units Other Than Participants: composite fillings
Arm/Group | Standard Care | Plasma Treatment
Number analyzed (Participants) | 27 | 21
Number analyzed (composite fillings) | 67 | 54
composite fillings | 2 | 0

ADVERSE EVENTS:
Arm/Group | Standard Care | Plasma Treatment
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/47
Other Adverse Events (participants affected / at risk) | 0/55 | 0/47

LIMITATIONS AND CAVEATS:
No limitation is reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No